CLINICAL TRIAL: NCT05350306
Title: Evaluation of the Dimensional Changes in the Mandible, Condyles, and the Temporomandibular Joint Following Skeletal Class III Treatment With the Chin Cup Using Low-Dose Computed Tomography
Brief Title: The Effects of the Chin Cup on Temporomandibular Joint and Mandibular Dimensions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-09-2022
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Class III Malocclusion
Keywords: chin cup; low-dose computed tomography; condyle-mandibular dimensions
MeSH Terms: conditions — Malocclusion, Angle Class III | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chincup (Experimental): Patients will be treated with occipital chincup and bonded bite block.
  Interventions: Device: Chincup
- Untreated subjects (Active Comparator): Patients will not undergone any treatment for 16 months.
  Interventions: Other: Control group

INTERVENTIONS:
Device: Chincup — Patients will receive an individual fabricated bonded bite block and occipital chincup. A 400-500g/side retroactive force will be applied in the direction of the condyles. Patients or panthers will be instructed to wear the appliance /14-16/ hours a day.
  Arms: Chincup
Other: Control group — The changes in condyle-mandibular volumes and superficial areas and relative positions of the condyles and glenoid fossa will be calculated after 16 months of observation.
  Arms: Untreated subjects

SUMMARY:
This in vivo comparative study will evaluate the changes in the mandibular dimensions and the glenoid fossa after skeletal class III subjects' therapy by chincup appliance and compare it with an untreated class III control group. Pre and post-treatment low-dose computed tomography images will be taken before and after achieving positive overjet and undergoing 16 months of active treatment/ observation. Dimensional and volumetric changes in the mandible, condyles, and glenoid fossa will be calculated and compared to those observed in the control group.

DETAILED DESCRIPTION:
Chincup is a usual treatment strategy for growing subjects with skeletal Class III malocclusions due to the mandibular overgrowth. However, the review of the literature reveals controversies and contradictions regarding the efficacy of chincup therapy in the retardation of mandibular growth. Moreover, the adaption of the temporomandibular joint (TMJ) following this treatment isn't clear yet. Two recent systematic reviews recommended the need for high-quality studies.

Computed tomography has been considered an ideal tool for evaluating the TMJ with the possibility of determining the real dimensions of the structures under study. Low-dose computed tomography was introduced as an alternative procedure with an effective dose proximately equal to traditional radiographs. Moreover, the volumetric analysis afforded by 3D imaging has proven reliable and accurate in the evaluation of mandibular and condylar sizes. Therefore, the objective of this randomized control trial is to evaluate the dimensional changes in the mandible, condyles, and glenoid fossa after chin cup therapy for children with mandibular prognathism in comparison with untreated Class III patients

Methods: patients ages between 6 and 8 with anterior crossbite, Class III relationships of the permanent first molars or mesial step relationships of the primary second molars, and short-faced pattern, will be selected from the orthodontic department in the faculty of dentistry at Damascus university. Thirty-eight subjects will be enrolled on the study, who will meet the following radiological inclusion criteria based on cephalometric images: Mild to moderate skeletal class III (4- <the sagittal skeletal angle< 0 degree), due to mandibular protrusion (SNB > 80°), and normal or horizontal growth pattern (Bjork's sum ≤396° ±5°).

Patients in the experimental group will receive an individual fabricated bonded bite block and occipital chincup. A 400-500g/side retroactive force will be applied in the direction of the condyles. Patients or panthers will be instructed to wear the appliance /14-16/ hours a day. Pre-(T1) and post-treatment (T2) low-dose computed tomography images will be taken after a positive overjet of 2-4 mm is obtained and undergoing 16 months of active treatment/ observation. The changes in condyle-mandibular volumes and superficial areas and relative positions of the condyles and glenoid fossa will be calculated and compared with those of untreated. Statistical analysis will be done by using the Statistical Package for Social Sciences, Windows version 26.0 (SPSS Inc., Chicago, Illinois, USA) Paired t-test and Wilcoxon signed-rank tests will be used for intragroup comparisons. For the intergroup comparisons, independent t-tests and Mann-Whitney U tests will be carried out.The confidence level is 95% (P< 0.05).

ELIGIBILITY:
Inclusion Criteria:

Clinical Inclusion criteria:

1. Children ages 6-8 years with anterior crossbite or edge-to-edge incisor relationship.
2. Class III relationships of the permanent first molars or mesial step relationships of the primary second molars.
3. the absence of centric relation and maximum intercuspation discrepancy
4. short-face pattern, adequate overbite.

Radiological Inclusion criteria:

1. Mild to moderate skeletal class III (4- <the sagittal skeletal angle (ANB)< 0 degree), due to mandibular protrusion (SNB > 80°).
2. normal or horizontal growth pattern (Bjork's sum ≤396° ±5°)

Exclusion Criteria:

1. temporomandibular joint disorders
2. craniofacial anomalies
3. history of previous orthodontic treatment

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in the mandibular volume and superficial area | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  After a semiautomatic segmentation will be utilized to isolate the mandibular bone, the mandible will be rendered in high-quality 3D model. Then, the crowns of the teeth will be removed by a plane passing through 1 mm inferior to the alveolar bone and 10 mm distal to the second primary molars. The mandible volumes and surface sizes will be automatically calculated by the software in mm3 and mm2, respectively.
Changes in the condylar volume and superficial area | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The condyles will be cut from 3D rendered mandibular model at neck level using a plane parallel to the Frankfort horizontal plane at the most inferior part of the sigmoid notch, the condyle volumes and surface sizes will be automatically calculated by the software in mm3 and mm2, respectively.
Change in the mandibular body (Go-Gn) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  Distance between the Gonion point and the Gnathion point.
Change in the ramus height (Co-Go) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  Distance between the Condylion point and the Gonion point.
Change in the total body length (Co-Gn) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  Distance between the Condylion point and the Gnathion point.
Change in the mandibular angle (GN-Go-CO) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The angle between the Condylion point, the Gonion point and Gnathion point.
Change in the vertical position of the condyle (CP-FH) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The measurement will be made on the corrected sagittal view: Distance of Condylar posterior point from Frankfort horizontal plane.
Change in the sagittal position of the condyle (CP-Y) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The measurement will be made on the corrected sagittal view: Distance of Condylar posterior point from Perpendicular plane (Y).
change in the vertical position of the mandibular fossa (FP-FH) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The measurement will be made on the corrected sagittal view: Distance of Fossa posterior point from Frankfort horizontal plane (FH).
Change in the sagittal position of the mandibular fossa (FP-Y) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The measurement will be made on the corrected sagittal view: Distance of point Fossa posterior point from Perpendicular plane (Y).
Quantitative changes of displacement of superimposed 3D mode | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The T1 and T2 3D volumes will be superimposed manually followed by automatic global registration. The point-based analysis will be performed to assess the changes in 3D mandibular models between T1 and T2, and a colour map will be produced. Quantitative mean, minimum, and maximum values of part analyses will be reported for comparative analyses.

SECONDARY OUTCOMES:
Change in the anterior joint space (AJS) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The measurement will be made on the corrected sagittal view: Distance between Condylar anterior point and Fossa anterior point.
Chang in the superior joint space (SJS) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The measurements will be made on the corrected sagittal view: Distance between Condylar posterior point and Fossa superior point.
Chang in the posterior joint space (PJS) | (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment
  The measurements will be made on the corrected sagittal view: Distance between Condylar posterior point and Fossa posterior point.

CONTACTS AND LOCATIONS:
Overall Officials: Amr H Husson, DDS,MSc,PhD, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y Hajeer, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria; Ahamd S Burhan, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria; Fehmieh R Nawaya, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chatzoudi MI, Ioannidou-Marathiotou I, Papadopoulos MA. Clinical effectiveness of chin cup treatment for the management of Class III malocclusion in pre-pubertal patients: a systematic review and meta-analysis. Prog Orthod. 2014 Dec 2;15(1):62. doi: 10.1186/s40510-014-0062-9. PMID 25679781
- [Background] Liu ZP, Li CJ, Hu HK, Chen JW, Li F, Zou SJ. Efficacy of short-term chincup therapy for mandibular growth retardation in Class III malocclusion. Angle Orthod. 2011 Jan;81(1):162-68. doi: 10.2319/050510-244.1. PMID 20936970
- [Background] Zurfluh MA, Kloukos D, Patcas R, Eliades T. Effect of chin-cup treatment on the temporomandibular joint: a systematic review. Eur J Orthod. 2015 Jun;37(3):314-24. doi: 10.1093/ejo/cju048. Epub 2014 Sep 1. PMID 25179261
- [Background] Swennen GR, Schutyser F. Three-dimensional cephalometry: spiral multi-slice vs cone-beam computed tomography. Am J Orthod Dentofacial Orthop. 2006 Sep;130(3):410-6. doi: 10.1016/j.ajodo.2005.11.035. PMID 16979502
- [Background] Lo Giudice A, Ronsivalle V, Grippaudo C, Lucchese A, Muraglie S, Lagravere MO, Isola G. One Step before 3D Printing-Evaluation of Imaging Software Accuracy for 3-Dimensional Analysis of the Mandible: A Comparative Study Using a Surface-to-Surface Matching Technique. Materials (Basel). 2020 Jun 21;13(12):2798. doi: 10.3390/ma13122798. PMID 32575875
- [Background] Cordasco G, Portelli M, Militi A, Nucera R, Lo Giudice A, Gatto E, Lucchese A. Low-dose protocol of the spiral CT in orthodontics: comparative evaluation of entrance skin dose with traditional X-ray techniques. Prog Orthod. 2013 Sep 10;14:24. doi: 10.1186/2196-1042-14-24. PMID 24325970
- [Background] Ikeda K, Kawamura A. Assessment of optimal condylar position with limited cone-beam computed tomography. Am J Orthod Dentofacial Orthop. 2009 Apr;135(4):495-501. doi: 10.1016/j.ajodo.2007.05.021. PMID 19361736
- [Derived] Husson AH, Burhan AS, Hajeer MY, Nawaya FR. Evaluation of the dimensional changes in the mandible, condyles, and the temporomandibular joint following skeletal class III treatment with chin cup and bonded maxillary bite block using low-dose computed tomography: A single-center, randomized controlled trial. F1000Res. 2023 Mar 13;12:264. doi: 10.12688/f1000research.130941.1. eCollection 2023. PMID 37008891